CLINICAL TRIAL: NCT03428061
Title: The ZWOlle Transmural Integrated Care for CArdiovaScular Risk Management Study
Acronym: ZWOT-CASE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: UMC Utrecht (Other)
Collaborators: Isala (Other); Medrie Health Care Group, Zwolle (Unknown); Hein Hogerzeil Stichting (Unknown)
Responsible Party: Principal Investigator, Monika Hollander, MD, PhD, MD PhD, UMC Utrecht
Other Study IDs: 57867
Record Dates: First submitted 2018-01-26; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Diseases; Hypercholesterolemia; Hypertension
Keywords: Prevention; Disease Management; Integrated care; Primary Health Care
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: The intervention under study will be the integrated care for cardiovascular risk management (CVRM), based on the Dutch CVRM guideline. Patients with a history of cardiovascular disease (CVD), a high cardiovascular risk (CVR) (>10%) or use of antihypertensives or lipid lowering drugs are included in the program. Patients will be invited for an intake consultation, including a blood test, an interview, physical examination and estimation of the 10-years cardiovascular risk. If indicated, treatment with medication will be started and general lifestyle advises will be given. Patients can be referred to smoking cessation therapy, dietician and exercise programs or a physiotherapist. Patients will be controlled on a regular base to evaluate and adjust their personal goals.
  Interventions: Other: Integrated care for cardiovascular risk management
- Control group: Usual care will be based on the Dutch CVRM guideline, describing how to calculate the CVR and advices to lower this risk by lifestyle intervention and/or medication. However systematic identification of patients eligible for CVRM, actively inviting patients for a visit, regular follow-up and standardized collaboration with other disciplines in the health care chain are not necessarily part of usual care.

INTERVENTIONS:
Other: Integrated care for cardiovascular risk management — Disease management program for the prevention of cardiovascular diseases
  Groups: Intervention group

SUMMARY:
Cardiovascular disease (CVD) contributes importantly to mortality and morbidity. Prevention of CVD by lifestyle change and medication is important and needs full attention.

In the Netherlands an integrated program for cardiovascular risk management (CVRM), based on the Chronic Care Model (CCM), has been introduced in many regions in recent years, but evidence from studies that this approach is beneficial is very limited.

In the ZWOT-CASE study the investigators will assess the effect of integrated care for CVRM in the region of Zwolle on two major cardiovascular risk factors: systolic blood pressure (SBP) and low-density lipoprotein cholesterol (LDL-cholesterol) in patients with or at high risk of CVD.

This study is a pragmatic clinical trial comparing integrated care for CVRM with usual care among patients aged 40-80 years with CVD (n= 370) or with a high CVD risk (n= 370) within 26 general practices. After one year follow-up, primary outcomes (SBP and LDL-cholesterol level) are measured. Secondary outcomes include lifestyle habits (smoking, dietary habits, alcohol use, physical activity), risk factor awareness, 10-year risk of cardiovascular morbidity or mortality, health care consumption, patient satisfaction and quality of life.

ELIGIBILITY:
Inclusion criteria for patients with CVD:

* Patients with a history of atherosclerotic CVD defined as documented angina pectoris, myocardial infarction, chronic ischemic heart disease, coronary sclerosis, transient ischaemic attack (TIA), cerebral infarction, intermittent claudication or aneurysm of the abdominal aorta
* The CV risk of the patient is managed in primary care, not in the hospital or outpatient clinic by a medical specialist
* Age between 40 and 80 years

Inclusion criteria for high risk patients:

* Use of blood pressure lowering or lipid lowering drugs
* A 10 -years CV risk > 10%, based on the Dutch guideline for CVRM and i) either 1 strongly cardiovascular risk enhancing factor or 2 mildly cardiovascular risk enhancing factors (see table 6) or ii) > 1 CV risk factor (current smoking, SBP>140 mmHg, LDL>2.5 mmol/L, TC/HDL-ratio > 8, chronic renal impairment (age < 65 years: eGFR < 60 ml/min/1,73 m2; age ≥ 65 years: eGFR < 45 ml/min/1,73 m2, and/or (micro)albuminuria).
* A 10-year CV risk of >20% and > 1 CV risk factor (current smoking, SBP>140 mmHg, LDL>2.5 mmol/L, TC/HDL-ratio > 8, chronic renal impairment (age < 65 years: eGFR < 60 ml/min/1,73 m2; age ≥ 65 years: eGFR < 45 ml/min/1,73 m2, and/or (micro)albuminuria).
* The CV risk of the patient is managed in primary care, not in the hospital or outpatient clinic by a medical specialist
* Age between 40 and 80 years

Exclusion criteria for all patients:

* Diabetes mellitus, as these patients are already included in a disease management program for diabetes mellitus
* Limited life expectancy, as assessed by the GP
* Cognitive impairment, as assessed by the GP
* No Dutch language proficiency
* Staying abroad for longer than three months during the duration of the study.
* The CV risk of the patient is managed in the hospital or outpatient clinic by a medical specialist

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The ZWOT-CASE study population will consist of a subgroup of 370 patients from the integrated CVRM care group (intervention) and 370 patients in the usual care (control) group. Both groups consist of respectively i) 185 patients with known CVD and ii) 185 patients with a high (>10%) ten year risk of CVD morbidity and mortality based on the Dutch Guideline for CVRM.
Sampling Method: Non-Probability Sample
Enrollment: 740 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | After 1 year of follow-up
  Systolic blood pressure, manual or electronic oscillometric measurement, at least 2 measurements with an interval of 1-2 minutes
LDL-cholesterol | After 1 year of follow-up
  Blood sample

SECONDARY OUTCOMES:
10-years cardiovascular morbidity or mortality risk | After 1 year of follow-up
  10-years cardiovascular morbidity or mortality risk (percentage) (Risk chart Dutch guideline or SMART risk score)
Smoking status | After 1 year of follow-up
  Smoking yes or no
Body mass index (BMI) | After 1 year of follow-up
  The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms and height in metres. BMI will be measured by the general practitioner or practice nurse during the endpoint visit
Healthy diet | After 1 year of follow-up
  Healthy diet yes or no according to the Dutch guideline for cardiovascular risk management and national guideline for healthy diet ((daily 150 - 200 grams vegetables and 200 grams fruit; daily 30 - 40 grams dietary fibers; twice a week 100 - 150 gram fish, at least once fatty fish; maximum of 6 grams salt per day; maximum of 2 (men) or 1 (women) alcohol consumptions per day). Food habits will be measured by a questionairre.
Physical activity | After 1 year of follow-up
  Squash questionnaire
Motivation to quit smoking | After 1 year of follow-up
  Motivation to quit smoking: motivated to quit/not motivated to quit/ considers to quit smoking
Awareness of received lifestyle advices | After 1 year of follow-up
  Aware/ not aware of received lifestyle advices, measured by questionairre
Awareness of food habits | After 1 year of follow-up
  Patient will be asked whether he/she thinks if he/she has healthy food habits yes or no. Measured by a questionairre
Awareness of physical activity | After 1 year of follow-up
  Patient will be asked whether he/she thinks if he/she has a healthy level of physical activity yes or no. Measured by a questionairre
Awareness of weight | After 1 year of follow-up
  Patient will be asked whether he/she thinks if he/she has a healthy weight yes or no. Measured by a questionairre
Awareness of hyperlipidaemia | After 1 year of follow-up
  Patient will be asked whether he/she thinks if he/she has hyperlipidaemia yes or no. Measured by a questionairre
Awareness of cardiovascular disease risk | After 1 year of follow-up
  Estimation by patient of his/her own cardiovascular disease risk by a questionairre
Awareness of hypertension | After 1 year of follow-up
  Patient will be asked whether he/she thinks if he/she has hypertension yes or no. Measured by a questionairre
Use of adequate antihypertensives | After 1 year of follow-up
  Use of adequate antihypertensives according to Dutch guideline for cardiovascular risk management. Measured by medication registered in electronic medical records in general practice
Use of adequate lipid lowering drugs | After 1 year of follow-up
  Use of adequate lipid lowering drugs according to Dutch guideline for cardiovascular risk management. Measured by medication registered in electronic medical records in general practice
Use of adequate anticoagulants | After 1 year of follow-up
  Use of adequate anticoagulants according to Dutch guideline for cardiovascular risk management. Measured by medication registered in electronic medical records in general practice
Morbidity | After 1 year of follow-up
  Newly developed cardiovascular diseases
Newly developed diabetes mellitus | After 1 year of follow-up
  Newly developed diabetes mellitus, based on coded diagnosis in electronic medical record in general practice
Newly developed COPD | After 1 year of follow-up
  Newly developed COPD, based on coded diagnosis in electronic medical record in general practice
Newly developed heart failure | After 1 year of follow-up
  Newly developed heart failure, based on coded diagnosis in electronic medical record in general practice
Newly developed atrial fibrillation | After 1 year of follow-up
  Newly developed atrial fibrillation, based on coded diagnosis in electronic medical record in general practice
Mortality | After 1 year of follow-up
  Died due to cardiovascular disease or other cause
Primary treating practitioner in the context of cardiovascular risk management | After 1 year of follow-up
  General practitioner or medical specialist.
Health care consumption in the past year | After 1 year of follow-up
  Consultations in the contect ox cardiovascular risk management in general practice
Self-management in the past year | After 1 year of follow-up
  Patient Activity Measure (PAM)
Self-measurements of blood pressure in the past year | After 1 year of follow-up
  Self-measurements of blood pressure in the past year yes or no
Patient satisfaction regarding the provided care in the past year | After 1 year of follow-up
  Patient Reported Experience Measure (PREM)
Quality of life | After 1 year of follow-up
  EQ-5D
Quality of life | After 1 year of follow-up
  SF-12
Anxiety and depression | After 1 year of follow-up
  Hospital Anxiety and Depression Scale (HADS), 0-7: no depression or anxiety, 8-10: depression or anxiety is possible,11-21: depression or anxiety is likely
Cost-efficiency | After 1 year of follow-up
  iPCQ

CONTACTS AND LOCATIONS:
Overall Officials: Arno Hoes, Prof. MD PhD, Study Chair — Julius Center for Health Sciences and Primary Care/ University Medical Center Utrecht; Monika Hollander, MD PhD, Principal Investigator — Julius Center for Health Sciences and Primary Care/ University Medical Center Utrecht; Arnoud van 't Hof, Prof. MD PhD, Principal Investigator — Maastricht University Medical Center, department of cardiology
Locations (1):
- General Practices, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM. [2016 European guidelines on cardiovascular disease prevention in clinical practice. The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts. Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation]. G Ital Cardiol (Rome). 2017 Jul-Aug;18(7):547-612. doi: 10.1714/2729.27821. No abstract available. Italian. PMID 28714997
- [Result] Dyakova M, Shantikumar S, Colquitt JL, Drew CM, Sime M, MacIver J, Wright N, Clarke A, Rees K. Systematic versus opportunistic risk assessment for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2016 Jan 29;2016(1):CD010411. doi: 10.1002/14651858.CD010411.pub2. PMID 26824223
- [Result] Khunti K, Stone M, Paul S, Baines J, Gisborne L, Farooqi A, Luan X, Squire I. Disease management programme for secondary prevention of coronary heart disease and heart failure in primary care: a cluster randomised controlled trial. Heart. 2007 Nov;93(11):1398-405. doi: 10.1136/hrt.2006.106955. Epub 2007 Feb 19. PMID 17309907
- [Result] Ebrahim S, Taylor F, Ward K, Beswick A, Burke M, Davey Smith G. Multiple risk factor interventions for primary prevention of coronary heart disease. Cochrane Database Syst Rev. 2011 Jan 19;2011(1):CD001561. doi: 10.1002/14651858.CD001561.pub3. PMID 21249647
- [Derived] Marchal S, Hollander M, Schoenmakers M, Schouwink M, Timmer JR, Bilo HJG, Schwantje O, van 't Hof AWJ, Hoes AW. Design of the ZWOT-CASE study: an observational study on the effectiveness of an integrated programme for cardiovascular risk management compared to usual care in general practice. BMC Fam Pract. 2019 Nov 1;20(1):149. doi: 10.1186/s12875-019-1039-z. PMID 31675925